CLINICAL TRIAL: NCT06121778
Title: Maintien A Domicile de la Personne âgée : évaluation Des déterminants Intra- extrinsèques Qui MAXimisent Cette possibilité
Brief Title: Home Support for Elderly: Evaluation of Intra- Extrinsic Determinants Which Maximize This Possibility
Acronym: MADMAX
Status: Not yet recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: 2022/7111
Record Dates: First submitted 2023-10-27; First posted 2023-11-08 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-06

CONDITIONS: Aging; Functional Disturbance; Home
MeSH Terms: interventions — Home Care Services

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Home: Elderly people living at home
  Interventions: Other: Home

INTERVENTIONS:
Other: Home — There is no intervention but evaluations of elderly persons living at home will be conducted every three years and for the next 12 years. If some people leave the home, as far as possible, the reason will be asked.

SUMMARY:
The French National Institute of Statistics and Economic Studies (INSEE) projects that the number of people aged 75 and over will increase in France from 5.2 million in 2007 to 11.6 million in 2060 (i.e., a 123% increase) and that of those aged 85 and over 1.3 to 5.4 million (315% increase). The marked increase in this segment of the population poses numerous practical and ethical questions regarding adaptation to our society, particularly in terms of medico-social offers. More specifically, surveys carried out among French people show an important paradox: almost 90% of those questioned want to be able to age in their home, but at the same time only a small part (estimated at 6%) of the French homes is adapted to the aging of its population. This inconsistency places the question of housing at the center of current public policies.

If current societal concerns raise the question of need to find alternatives to entering an institution, a research work addressing all dimensions impacted by life at home for the elderly (quality of life, maintenance of functional, decision-making skills, nutritional status, etc.) jointly in the same population area and at different times (i.e., until leaving home for some people) remains to be carried out to allow us to better understand the nature and functioning of these factors, and thus propose integrated models. Indeed, too often these questions are studied separately on different populations and at different stages different from the life of the elderly person. Unfortunately, this does not allow us to clearly perceive the importance specificity takes on each factor, nor whether the proposals made really meet the objectives assigned to them. These questions relate in particular to: what aspects related to the person or their environment they contribute, when the person wishes, to be able to stay and live in your home? Since the departure of domicile would be postponed, does this mean that it is carried out due to the state health of the elderly worse? Understanding the relationship between the elderly and their housing will make it possible to draw up an inventory of the premises necessary for construction of the steps which will follow and which will be carried out by the different partners, in particular the public authorities, associations, social landlords (e.g., implementation of new clinical studies, health promotion, policy support, urban and housing planning, etc.). As part of an action-research program (concrete actions and transformative in the field), and relying on the approaches already underway, the main objective of this project will be to determine in elderly people living at home independent what are the main intrinsic factors and extrinsic elements that allow/promote this way of life.

ELIGIBILITY:
Inclusion Criteria:

* Men and women living at home alone, as a couple or accompanied (children, relatives, etc.). For people living as a couple, if both meet all the criteria, both members of the couple can be evaluated; Being between 70 and 75 years old; Independent people physically capable of moving around (Iso Ressource Group [GIR] 5 and 6); GIR 5 includes people moving around alone within their home, eating and dressing alone. They may need occasional help with washing and domestic activities (meal preparation, cleaning, etc.); GIR 6 is made up of people who are autonomous for all discriminatory acts of everyday life. They may need occasional help with domestic activities; Living in a primary residence in Franche Comté region; Not objecting to participation in the study; Being affiliated to a French social security scheme or beneficiary of such a scheme.

Exclusion Criteria:

* Having made a request for living in an alternative hose or waiting for a response; Having an episode of acute pathology; Having major cognitive impairment (assessed using the Mini Mental State Examination [MMSE] and a threshold > 20 [mild or no impairment]) (23); Having a contraindication to physical exercise; Having artificial nutrition or having replacement treatment (e.g. dialysis); Being legally incapacitated or in limited legal capacity; Person unlikely to cooperate in the study and/or low cooperation anticipated by the investigator; Not expressing himself easily in French.

Ages: 70 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Independent elderly people living in the region of Franche-Comté (France).
Sampling Method: Probability Sample
Enrollment: 274 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2023-11-01 (Estimated); Study Completion 2035-10-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of elderly people remained at home (%) | 12 years
  To determine the percentage of elderly people who remained at home at the end of the project (after 12 years) and their characteristics.

IPD SHARING:
Plan to Share IPD: No